CLINICAL TRIAL: NCT00758329
Title: Retrospective Data Review of ReCap Total Hip Resurfacing
Status: Withdrawn | Type: Observational
Why Stopped: No further contact with the site
Sponsor: Zimmer Biomet (Industry)
Collaborators: Biomet U.K. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: BMET UK 09
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Osteoarthritis of the Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Device: ReCap Total Hip Resurfacing

INTERVENTIONS:
Device: ReCap Total Hip Resurfacing — ReCap Total Hip Resurfacing

SUMMARY:
Retrospective Data Review on clinical outcomes and survivorship of ReCap Total Hip Resurfacing

ELIGIBILITY:
Inclusion:

* Patients received ReCap total hip resurfacing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received ReCap Total Hip Resurfacing
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2004-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Survival rate | 2 yr

SECONDARY OUTCOMES:
Harris Hip Score | 2yr